CLINICAL TRIAL: NCT04983186
Title: mBrain-21 : a Three-month Study on Context-awareness, Physiological Monitoring, and Machine Learning in Migraine and Cluster Headache
Acronym: MBRAIN-21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BC-10031
Record Dates: First submitted 2021-07-05; First posted 2021-07-30 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Migraine; Cluster Headache
Keywords: Migraine; Cluster Headache; Smartphone application; Machine Learning; Wearable sensor
MeSH Terms: conditions — Migraine Disorders; Cluster Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Participants wear the Empatica E4 wearable sensor and use the smartphone applications developed by the research team.
  Interventions: Device: Wearable sensor and smartphone application

INTERVENTIONS:
Device: Wearable sensor and smartphone application — Empatica E4 wearable sensor and custom-made headache smartphone application

SUMMARY:
This study collects data from migraine and cluster headache patients during a three-month study. Contextual data (e.g. location or smartphone usage) and physiological variables will be used to assist machine learning algorithms in making predictions on activity, stress and sleep in patients with migraine or cluster headache.

DETAILED DESCRIPTION:
Migraine and cluster headache are brain disorders with disabling headache attacks and assoicated symptoms. Attacks have multiple phases such as the premonitory phase, aura phase, headache phase and postdromal phase. During those phases, symptoms of homeostatic disturbance or sensory alterations may occur.

The goal of the study is to observe activity, stress and sleep parameters in relation to registered headache attacks.

Participation in the mBrain-21 study will last maximum 90 days. Participants are patients with migraine or cluster heacache recruited within the headache clinic of Ghent University Hospital. Physiological variables such as heart rate, movement and galvanic skin resonse will be measured by the Empatica E4 wrist sensor. Patient-specific experiences during headache attacks and activities of daily life will be registered with a custom-made headache smartphone applications. Contextual data (e.g. smartphone usage or location) can be autonomously collected through smartphone applications.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants between the age of 18 en 65 years.
* Diagnosis of migraine without aura (ICHD-3 diagnosis 1.1) or migraine with aura (ICHD-3 diagnosis 1.2) or chronic migraine (ICHD-3 diagnosis 1.3)
* Headache crystal clear days on minimum 5 days per month on average.
* Onset of headache syndrome before the age of 50.
* Attacks of migraine or cluster headache are clearly distinguishable from other types of headache disorders if present.
* Participant complies with protocol to use smartphone applications on his or her own Android-based smartphone (minimum version 8.0) and to provide access to his or her smartphone dataplan.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Accuracy (F1-scores) machine learning algorithms | After 90 days
  Machine learning algorithms for stress detection, sleep detection, activity detection and headache attack detection

SECONDARY OUTCOMES:
Demographics | At the beginning of the study
  Demographic characteristics of participants
Headache phenotype characteristics | At the beginning of the study
  Headache phenotype characteristics
Migraine Specific Questionnaire v2.1 | After 90 days
  Migraine Specific Questionnaire v2.1
MIDAS Migraine Disability Assessment | After 90 days
  MIDAS Migraine Disability Assessment
MOS Short-Form General Health Survey (SF-20) | After 90 days
  MOS Short-Form General Health Survey (SF-20)
Pittsburgh Sleep Quality index | After 90 days
  Pittsburgh Sleep Quality index
MUltilevel Assessment of Interoceptive Awareness v2 (MAIAv2) | After 90 days
  MUltilevel Assessment of Interoceptive Awareness v2 (MAIAv2)
Perceived Stress Scale (PSS-10) | After 90 days
  Perceived Stress Scale (PSS-10)
Connor Davidson Resilience Scale (CD-RISC 25) | After 90 days
  Connor Davidson Resilience Scale (CD-RISC 25)
Penn State Worry Questionnaire (PSWQ) | After 90 days
  Penn State Worry Questionnaire (PSWQ)
Perseverative Thinking Questionnaire (PTQ) | After 90 days
  Perseverative Thinking Questionnaire (PTQ)
Ruminative Response Scale (RRS) | After 90 days
  Ruminative Response Scale (RRS)
Basic Needs Scale | After 90 days
  Basic Needs Scale
Emotion Regulation Scale | After 90 days
  Emotion Regulation Scale
Neuroticism (subscale from BFI) | After 90 days
  Neuroticism (subscale from BFI)

OTHER OUTCOMES:
Feedback from participants | After 90 days
  Feedback from participants on compliance, adherence, usability and user experience of study infrastructure

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Ghent: Department of Neurology, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Van Der Donckt J, Vandenbussche N, De Brouwer M, Steenwinckel B, Stojchevska M, Ongenae F, Paemeleire K, Van Hoecke S. Analysis of free-living daytime movement in patients with migraine with access to acute treatment. J Headache Pain. 2025 Feb 13;26(1):33. doi: 10.1186/s10194-025-01971-y. PMID 39948510